CLINICAL TRIAL: NCT03071757
Title: A Multicenter, Phase 1, Open-Label, Dose-Escalation Study of the Safety, Tolerability and Pharmacokinetics of ABBV-368 as a Single Agent and Combination in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of the Safety, Tolerability and Pharmacokinetics of ABBV-368 as a Single Agent and Combination in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-074; 2016-004205-14 (EudraCT Number)
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Solid Tumors; Cancer; Metastatic Solid Tumors; Advanced Solid Tumors; Triple negative breast cancer (TNBC); Ovarian cancer; Hepatocellular carcinoma (HCC); Gastric cancer; Mesothelioma; Small cell lung cancer (SCLC); Cholangiocarcinoma; Merkel cell carcinoma; Melanoma; Non-small cell lung cancer (NSCLC); 2'-Deoxy-2'-[18F]Fluoro-9-β-DArabinofuranosylguanine (18F-AraG)
MeSH Terms: conditions — Neoplasms; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Carcinoma, Hepatocellular; Stomach Neoplasms; Mesothelioma; Small Cell Lung Carcinoma; Cholangiocarcinoma; Carcinoma, Merkel Cell; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1A: Monotherapy Dose Escalation (Experimental): Part 1A: ABBV-368 (various dose levels) intravenous administration every 2 weeks (Q2W). One cycle of treatment is 28 days, thus there will be 2 doses with ABBV-368 per cycle.
  Interventions: Drug: ABBV-368
- Part 2A: Monotherapy Cohort Expansion (Experimental): Part 2A: Additional participants (triple negative breast cancer [TNBC]) will be enrolled in a dose expansion cohort that will further evaluate ABBV-368 (various dose levels) intravenous administration Q4W.
  Interventions: Drug: ABBV-368
- Part 2B: Combination Therapy Cohort Expansion (Experimental): Part 2B: Additional participants (with Head and Neck carcinoma) will be enrolled in a dose expansion cohort that will further evaluate ABBV-368 (various dose levels) intravenous administration Q4W plus ABBV-181.
  Interventions: Drug: ABBV-368; Drug: ABBV-181
- Part 3A: 18F-AraG Imaging Substudy in TNBC Participants (Experimental): Part 3A: Additional participants (with TNBC) will be enrolled in 18F-AraG Imaging Substudy that will further evaluate ABBV-368 intravenous administration Q4W plus ABBV-181.
  Interventions: Drug: ABBV-368; Drug: ABBV-181
- Part 3B: 18F-AraG Imaging Substudy in HNSCC Participants (Experimental): Part 3B: Additional participants (with HNSCC) will be enrolled in 18F-AraG Imaging Substudy that will further evaluate ABBV-368 intravenous administration Q4W plus ABBV-181.
  Interventions: Drug: ABBV-368; Drug: ABBV-181

INTERVENTIONS:
Drug: ABBV-368 — Intravenous infusion
Drug: ABBV-181 — Intravenous infusion
  Arms: Part 2B: Combination Therapy Cohort Expansion; Part 3A: 18F-AraG Imaging Substudy in TNBC Participants; Part 3B: 18F-AraG Imaging Substudy in HNSCC Participants

SUMMARY:
The primary purpose of this Phase 1, open-label study is to evaluate the safety, pharmacokinetics, and preliminary efficacy of ABBV-368 as a monotherapy and in combination with ABBV-181 in participants with locally advanced or metastatic solid tumors. The study will consist of 3 parts: ABBV-368 dose escalation, ABBV-368 tumor-specific dose expansion (triple negative breast cancer [TNBC] cohort and head and neck cancer cohort) and 18F-AraG Imaging Substudy.

DETAILED DESCRIPTION:
Recruitment is closed in Part 1A; subjects are in maintenance

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologic or cytology diagnosis of a known immunogenic solid tumor, as described for Part 1 Dose Escalation and Part 2 Cohort Expansion:
* Part 1 Dose Escalation:
* Participants with advanced or metastatic solid tumors that have exhausted standard treatment for their incurable disease and for whom there is currently no programmed cell death 1 (PD-1)/ programmed cell death-ligand 1 (PD-L1) approved therapy, with immunogenic type tumors such as, but not limited to triple negative breast cancer (TNBC), ovarian cancer, small cell lung cancer, mesothelioma, and cholangiocarcinoma.
* Participants who are refractory to a PD-1/PD-L1 agent, with tumor types such as melanoma, NSCLC, platinum-pretreated head and neck cancer, second line bladder and RCC.
* Part 2A and 2B Cohort Expansion:
* 2A : TNBC ABBV-368 monotherapy cohorts: Subjects with locally advanced or metastatic TNBC that have exhausted standard treatment for their incurable disease.
* 2B : Head and Neck cohort: Participants with recurrent squamous cell head and neck carcinoma that are not candidates for curative treatment with local or systemic therapy, or metastatic (disseminated) head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, and larynx that is considered incurable by local therapies.
* Part 3A and 3B Imaging Substudy:
* 3A: Participants with locally advanced or metastatic TNBC that have exhausted standard treatment for their incurable disease and are treatment naïve to a PD-1/PD-L1 targeting agent.
* 3B: Participants with recurrent HNSCC that are not candidates for curative treatment with local or systemic therapy, or metastatic HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx that is considered incurable by local therapies. Participants must be treatment naïve to a PD-1/PD-L1 targeting agent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
* Participants must have immune-related Response Evaluation Criteria for Solid Tumors (iRECIST) evaluable or measurable disease in the PART 1 and measurable disease per iRECIST in PART 2
* Adequate bone marrow, kidney and liver function.

Exclusion Criteria:

* Received anticancer therapy including chemotherapy, immunotherapy, radiation therapy, biologic, herbal therapy, or any investigational therapy within a period of 21 days prior to the first dose of ABBV-368.
* Prior treatment with an OX40 targeting agent.
* has known uncontrolled metastases to the central nervous system (CNS).
* History of active autoimmune disorders and other conditions that compromise or impair the immune system.
* Confirmed positive test results for human immunodeficiency virus (HIV), or subjects with chronic or active hepatitis A, B or C. Subjects who have a history of hepatitis B or C who have documented cures after anti-viral therapy may be enrolled.
* Has received live vaccine within 28 days prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Terminal half-life (t1/2) of ABBV-368 | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  Terminal half-life of ABBV-368
Area under the serum concentration-time curve (AUC) of ABBV-368 | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  Area under the serum concentration-time curve of ABBV-368
Maximum tolerated dose (MTD) of ABBV-368 when administered as monotherapy or in combination with ABBV-181 | Up to 1 year
  The MTD of ABBV-368 when administered as monotherapy or as combination therapy with ABBV-181 will be determined during the dose escalation phase of the study.
Recommended Phase 2 dose (RPTD) for ABBV-368 when administered as monotherapy or as combination therapy with ABBV-181 | Up to 18 months
  Recommended Phase 2 dose (RPTD) for ABBV-368 when administered as monotherapy or as combination therapy with ABBV-181 will be established during the Dose expansion of the study
Time to Cmax (Tmax) of ABBV-368 | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  Time to Cmax of ABBV-368
Terminal phase elimination rate constant (β) of ABBV-368 | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  Terminal phase elimination rate constant of ABBV-368
Number of Participants With Adverse Events | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs/TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Maximum observed serum concentration (Cmax) of ABBV-368 | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  Maximum observed serum concentration of ABBV-368

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  ORR is defined as the proportion of subjects with a confirmed partial or complete response to the treatment.
Clinical benefit rate (CBR) | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  CBR defined as the proportion of subjects with a confirmed partial response (PR), complete response (CR), or stable disease.
Duration of Objective Response (DOR) | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  DOR defined as the time from the initial objective response to disease progression or death, whichever occurs first.
Progression-Free Survival (PFS) | Multiple time points in each cycle (each cycle is 28 days), throughout study completion, an average of 2 years, or participant becomes lost to follow up, or study termination
  PFS time is defined as the time from the first dose of study drug (Day 1) to disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (27):
- United States (10):
  - Moores Cancer Center at UC San Diego /ID# 201334, La Jolla, California
  - University of California, Davis Comprehensive Cancer Center /ID# 201342, Sacramento, California
  - Stanford University /ID# 206949, Stanford, California
  - Yale University /ID# 207895, New Haven, Connecticut
  - Carolina BioOncology Institute /ID# 160786, Huntersville, North Carolina
  - Greenville Hospital System /ID# 160785, Greenville, South Carolina
  - University of Texas Southwestern Medical Center /ID# 201934, Dallas, Texas
  - South Texas Accelerated Research Therapeutics /ID# 160788, San Antonio, Texas
  - University of Virginia /ID# 212895, Charlottesville, Virginia
  - Virginia Cancer Specialists - Fairfax /ID# 160787, Fairfax, Virginia
- France (4):
  - AP-HM - Hopital de la Timone /ID# 165036, Marseille, Bouches-du-Rhone
  - Centre Leon Berard /ID# 165037, Lyon, Rhone
  - Institut Gustave Roussy /ID# 165035, Villejuif, Val-de-Marne
  - Institut Curie /ID# 165038, Paris, Île-de-France Region
- Japan (2):
  - National Cancer Center Hospital East /ID# 214530, Kashiwa-shi, Chiba
  - National Cancer Center Hospital /ID# 214531, Chuo-ku, Tokyo
- Pan American Center for Oncology Trials, LLC /ID# 213809, Rio Piedras, Puerto Rico
- Spain (7):
  - Hospital Duran i Reynals /ID# 205997, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda /ID# 206973, Majadahonda, Madrid
  - CLINICA UNIVERSIDAD DE NAVARRA-Pamplona /ID# 208879, Pamplona, Navarre
  - Hospital General Universitario Gregorio Maranon /ID# 205999, Madrid
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 205996, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 211500, Madrid
  - Hospital Clinico Universitario de Valencia /ID# 211499, Valencia
- Taiwan (3):
  - National Cheng Kung University Hospital /ID# 164002, Tainan
  - National Taiwan University Hospital /ID# 164000, Taipei
  - Taipei Medical University Hospital /ID# 164001, Taipei

IPD SHARING:
Plan to Share IPD: No